CLINICAL TRIAL: NCT03995212
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of Oral CR845 in Patients With Primary Biliary Cholangitis (PBC) and Moderate-to-Severe Pruritus
Brief Title: Study to Evaluate the Safety and Efficacy of Oral CR845 (Difelikefalin) in Patients With Primary Biliary Cholangitis (PBC) and Moderate-to-Severe Pruritus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment due primarily to Covid-19
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR845-210401
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Cholestatic Pruritus
Keywords: Primary Biliary Cholangitis; Pruritus; CR845; Chronic Itch; difelikefalin; Itch; Itching; Generalized pruritus
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Pruritus | interventions — difelikefalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CR845 1.0 mg (Active Comparator): Oral CR845 1.0 mg tablet administered twice daily
  Interventions: Drug: CR845 1.0 mg
- Placebo (Placebo Comparator): Oral placebo tablet administered twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CR845 1.0 mg — Oral CR845 1.0 mg administered twice daily
  Other Names: CR845; Difelikefalin
  Arms: CR845 1.0 mg
Drug: Placebo — Oral Placebo administered twice daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of twice-daily (BID) oral CR845 1.0 mg in patients with PBC with moderate-to-severe pruritus. The study includes a 16-week Treatment Period.

DETAILED DESCRIPTION:
This study will consist of a Screening Visit, a 7-day Run-in Period, a 16-week Treatment Period, and a Follow-up Visit (approximately 7-10 days after the last dose of study drug). Informed consent will be obtained prior to performing any study-specific procedures.

The Screening Visit will occur within 7 to 28 days prior to randomization to assess eligibility.

Day 1 of the Treatment Period will be defined as the day of the administration of the first dose of study drug. If patients continue to meet all inclusion and no exclusion criteria at the end of the 7-day Run-in Period, they will be randomized in a 1:1 ratio to receive either placebo or CR845 tablets at a dose of 1.0 mg orally BID for 16 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

* Confirmed diagnosis of PBC;
* If currently taking ursodeoxycholic acid (UDCA), should be on stable dose for >12 weeks prior to screening and plan on continuing to take UDCA throughout the study;
* If previously taking UDCA, should have discontinued its use >12 weeks prior to screening;
* Self-reports experiencing daily or near-daily pruritus during the month prior to screening;
* Prior to randomization has a mean baseline WI-NRS score indicative of moderate to severe pruritus.

Key Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

* Presence of Child-Pugh Class C decompensated cirrhosis at screening;
* Itching secondary to biliary obstruction;
* History or presence of hepatocellular carcinoma, hepatic abscess, or acute portal vein thrombosis;
* Current placement on liver transplantation list with anticipated liver transplant during the course of the study or current Model for End-stage Liver Disease (MELD) score ≥15;
* Alanine aminotransferase or aspartate aminotransferase >5 × upper limit of normal at screening, or within 2 months prior to screening;
* Anticipates receiving an opioid antagonist (eg, naloxone, naltrexone) or opioid-mixed agonist-antagonist (eg, buprenorphine, nalbuphine) from the start of screening through the end of the Treatment Period;
* New or change of treatment with antihistamines and corticosteroids (oral, intravenous, or topical), opioids, gabapentin, pregabalin, cholestyramine, rifampicin or fibrates within 14 days prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 16 with respect to the weekly mean of the daily 24-hour Worst Itching Intensity Numeric Rating Scale (WI-NRS) score. | Baseline, Week 16
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".

SECONDARY OUTCOMES:
Improvement in itch-related quality of life as assessed by the change from baseline to Week 16 in total Skindex-10 Scale score | Baseline, Week 16
  The Skindex-10 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: disease, mood/emotional distress, and social functioning domain. A lower total score represents better quality of life.
Improvement in itch-related quality of life as assessed by the change from baseline to Week 16 in 5-D Itch Scale score | Baseline, Week 16
  The 5-D Itch Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past 2 weeks. The questions cover five dimensions of itch including the degree, duration of itch/day, direction (improvement/worsening), disability (impact on activities such as work), and body distribution of itch. A lower total score represents better quality of life.
Reduction of itch intensity as assessed by the proportion of patients achieving an improvement from baseline ≥3 points with respect to the weekly mean of the daily 24-hour WI-NRS score at Week 16 | Week 16
  Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (14):
- United States (14):
  - Cara Therapeutics Study Site, Coronado, California
  - Cara Therapeutics Study Site, Rialto, California
  - Cara Therapeutics Study Site, San Francisco, California
  - Cara Therapeutics Study Site, Colorado Springs, Colorado
  - Cara Therapeutics Study Site, Miami, Florida
  - Cara Therapeutics Study Site, Plantation, Florida
  - Cara Therapeutics Study Site, Indianapolis, Indiana
  - Cara Therapeutics Study Site 2, Boston, Massachusetts
  - Cara Therapeutics Study Site, Boston, Massachusetts
  - Cara Therapeutics Study Site, New York, New York
  - Cara Therapeutics Study Site, Nashville, Tennessee
  - Cara Therapeutics Study Site, Arlington, Texas
  - Cara Therapeutics Study Site, Newport News, Virginia
  - Cara Therapeutics Study Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No